CLINICAL TRIAL: NCT06103201
Title: Utility of Hyperpolarized 13C-Pyruvate Metabolic Magnetic Resonance Imaging in the Diagnosis of Early Cerebral Metabolic Crisis After Traumatic Brain Injury
Brief Title: Hyperpolarized 13C-pyruvate Metabolic MRI With Traumatic Brain Injury
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jiachen Zhuo, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00104422
Record Dates: First submitted 2023-09-28; First posted 2023-10-26 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metabolic MRI in traumatic brain injury patients (Experimental): Perform metabolic magnetic resonance imaging on patients who have traumatic brain injury to understand early brain metabolism changes in this population
  Interventions: Drug: Hyperpolarized 13C-Pyruvate
- Metabolic MRI in subarachnoid hemorrhage patients (Experimental): Perform metabolic magnetic resonance imaging on patients who have subarachnoid hemorrhage to understand early brain metabolism changes in this population
  Interventions: Drug: Hyperpolarized 13C-Pyruvate
- Metabolic MRI in healthy volunteers (Experimental): Perform metabolic magnetic resonance imaging on healthy volunteers to understand early brain metabolism changes in this population
  Interventions: Drug: Hyperpolarized 13C-Pyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Hyperpolarized Pyruvate (13C) Injection, containing spin-polarized ("hyperpolarized") [13C]pyruvate, is being studied as a diagnostic agent in combination with 13C spectroscopic MR imaging. The aim is to visualize [13C]pyruvate and its metabolites and thereby distinguish between anatomical areas with normal vs. abnormal metabolism, which should be useful in diagnosing and characterizing, for example, traumatic brain injury.
  Hyperpolarized Pyruvate (13C) Injection and [13C]pyruvate are general terms used throughout this brochure, which refer to all 13C labeling patterns, such as [1- 13C]pyruvate, [2- 13C]pyruvate and [1,2- 13C]pyruvate. From biological and safety standpoints, pyruvate with each of the labeling patterns behaves identically in the human body [Koletzko et al., 1997].

SUMMARY:
The purpose of this study is to examine the safety and feasibility of using hyperpolarized metabolic MRI to study early brain metabolism changes in subjects presenting with head injury and suspected non-penetrating traumatic brain injury (TBI). This study will also compare HP pyruvate MRI-derived metrics in TBI patients with healthy subjects as well as Subarachnoid hemorrhage (SAH) patients to better understand if metabolic Magnetic resonance imaging scan (MRI) can improve our ability to diagnose a TBI.

The FDA is allowing the use of hyperpolarized [1-13C] pyruvate (HP 13C-pyruvate) in this study.

Up to 15 patients (5 with TBI, 5 with SAH, and 5 healthy volunteers) may take part in this study at the University of Maryland, Baltimore (UMB).

ELIGIBILITY:
Inclusion Criteria:

* History of acute head injury with or suspected non-penetrating acute TBI
* Suitable to undergo contrast-enhanced MRI
* Negative serum pregnancy test

Exclusion Criteria:

* Inability to undergo MRI scan
* Inability to receive IV MRI contrast agents secondary to severe reaction or renal insufficiency
* Positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
Measures of conversion of pyruvate to lactate (apparent conversion rate constant kPL, lactate-to-pyruvate ratio) and pyruvate to bicarbonate (apparent conversion rate constant kPB, bicarbonate-to-pyruvate ratio) | within two years post enrollment
  To assess the differences between the three patient groups

SECONDARY OUTCOMES:
Correlation of the conversion of pyruvate to lactate and pyruvate to bicarbonate measures with results from clinical and neuropsychological evaluation. | within two years post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Mayer, Dr. rer. nat., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States